CLINICAL TRIAL: NCT04348292
Title: A Phase 1b Neoadjuvant Trial of Sirolimus Followed by Durvalumab (MEDI4736) in Resectable Non-small Cell Lung Cancer
Brief Title: Sirolimus and Durvalumab for the Treatment of Stage I-IIIA Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual goal not met.
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Carlisle, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00116422; NCI-2019-07427 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4867-19 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH); P50CA217691 (NIH)
Record Dates: First submitted 2020-02-20; First posted 2020-04-16 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab; Immunoglobulin G; Disulfides; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sirolimus, durvalumab) (Experimental): Patients receive sirolimus PO QD on days 1-21 in the absence of disease progression or unacceptable toxicity. Starting on day 22, patients receive durvalumab IV over 1 hour. Treatment with durvalumab repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Within a 2-3 week period after the second dose of durvalumab, but not earlier than two weeks after the administration of durvalumab, patients undergo standard of care surgery.
  Interventions: Drug: Durvalumab; Drug: Sirolimus

INTERVENTIONS:
Drug: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217

SUMMARY:
This trial studies the side effects of sirolimus and durvalumab and to see how well they work in treating patients with stage I-IIIA non-small cell lung cancer. Sirolimus is an oral medication that blocks the mTOR cellular pathway which may help the immune system work better. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving sirolimus before durvalumab may help the immune system get rid of cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of sirolimus followed by durvalumab as neoadjuvant treatment II. To evaluate the efficacy of sirolimus followed by durvalumab as neoadjuvant treatment for stage I, II, and IIIA non-small cell lung cancer (NSCLC)

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of sirolimus in combination with durvalumab as neoadjuvant treatment for stage I, II, and IIIA NSCLC II. To evaluate response to sirolimus in combination with durvalumab in patients with PD-L1-positive versus (vs.) PD-L1-negative tumors III. To evaluate the association between blood mutation burden and response to sirolimus and durvalumab

EXPLORATORY OBJECTIVES:

I. To evaluate the immune-mediated effects of combination sirolimus and durvalumab II. To investigate tumor and immune microenvironment changes in tissue samples

OUTLINE:

Patients receive sirolimus orally (PO) once daily (QD) on days 1-21 in the absence of disease progression or unacceptable toxicity. Starting on day 22, patients receive durvalumab intravenously (IV) over 1 hour. Treatment with durvalumab repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Within a 2-3 week period after the second dose of durvalumab, but not earlier than two weeks after the administration of durvalumab, patients undergo standard of care surgery.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically documented NSCLC: Stage I, II, IIIa NSCLC based on 8th edition of American Joint Committee on Cancer (AJCC) Non-small cell Lung Cancer Staging system
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the United States [US]) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of >= 26 weeks
* Body weight > 30 kg
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) 1.5 x 10^9/L (>= 1500 per mm^3)
* Platelet count >= 100 x 10^9/L (>= 100,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be =< 5 x ULN
* Measured creatinine clearance (CL) > 40 mL/min or calculated creatinine CL > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Patients must consent to pre-treatment research biopsy and study peripheral blood collection
* Patients must have measurable disease, defined by RECIST v 1.1
* Patient is able to take oral medications
* Patient consents to heavy water (D2O) self-administration if on optional heavy water labelling study

Exclusion Criteria:

* Patients who have had prior therapy for lung cancer including chemotherapy, hormonal therapy, or radiotherapy
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study
* Prior treatment with anti-PD-1, anti-PDL-1, other PD-1/PDL-1 pathway targeting agents, or mTOR inhibition
* History of allogenic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for

  * Malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of investigational product (IP) and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* QT interval corrected for heart rate using Fridericia's formula (QTcF) >= 470 ms. Patient safety and the cardiac SKG should be consulted as needed
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment
* Patients with a history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Inability to stop prohibited concomitant medications
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer W Carlisle, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Sirolimus, Durvalumab)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: diagnosed with Resectable Non-small Cell Lung Cancer
Arm/Group | Treatment (Sirolimus, Durvalumab)
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (7.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v5.0
Description: Other adverse events will be listed and summarized by severity, seriousness, and by system organ class. The number and percentage of subjects who experience AEs will be presented in tabular and/or graphical format and summarized descriptively, where appropriate. The frequency of overall toxicity, categorized by toxicity grades 1 through 5, will be described.
Time Frame: at time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sirolimus, Durvalumab)
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Complete Pathologic Response
Description: Disappearance of all invasive cancer
Time Frame: at time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sirolimus, Durvalumab)
Number analyzed (Participants) | 2
Participants
  PDL-1 negative | 1
  PDL-1 positive | 1

3. Other Pre Specified Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: Any number of patients who experienced dose limiting toxicity
Time Frame: at time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sirolimus, Durvalumab)
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: adverse event data were collected from screening until surgical resection, an average of 12 weeks
Arm/Group | Treatment (Sirolimus, Durvalumab)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sirolimus, Durvalumab) (N=3)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
fatigue (General disorders) | 1 (1)
chyle leak (Blood and lymphatic system disorders) | 1 (1)
pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a low accruing trial which amassed fewer patients than anticipated. Due to stalled enrollment, the study was terminated and did not reach completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT04348292/Prot_SAP_000.pdf